CLINICAL TRIAL: NCT01083914
Title: Investigation of the Ability of the MECC System to Provide Reduced Risk Over the Existing CECC System and Equivalent Risk to Off-Pump CABG Surgery: The IMPROVE TRIAL
Brief Title: Comparing Blood Loss, RBC Transfusions and Inflammatory Marker Changes Among Methods of CPB
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 009-113
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease
Keywords: extracorporeal circulation, off-pump CABG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- OPCAB: Those who have CABG surgery off pump Those who have CABG surgery using conventional cardiopulmonary bypass Those who have CABG surgery using a minimal extracorporeal circulation system
- CPB: Those who have CABG surgery off pump Those who have CABG surgery using conventional cardiopulmonary bypass Those who have CABG surgery using a minimal extracorporeal circulation system
- MECC: Those who have CABG surgery off pump Those who have CABG surgery using conventional cardiopulmonary bypass Those who have CABG surgery using a minimal extracorporeal circulation system

SUMMARY:
The purpose of this study is to compare blood loss and the number of transfusions received by each patient having coronary bypass surgery. The second purpose is to determine how the level inflammation in patients during and after surgery may affect a patient's response to surgery and the recovery process.

DETAILED DESCRIPTION:
Off-pump coronary artery bypass grafting (OPCAB) and the use of minimal extracorporeal circulation system (MECC) have both been proposed as alternatives to avoid the harmful effects of conventional cardiopulmonary bypass (CPB). However, with the technically more demanding nature of off-pump CABG, the potential short-term benefits of off-pump surgery may not translate into long-term benefits in providing optimal revascularization. In this prospective cohort study, it is our goal to evaluate short term outcomes as demonstrated by blood loss, transfusion need, and systemic inflammatory response during CABG surgery using MECC or conventional CPB or OPCAB.

In addition to the technical challenges posed during off-pump CABG surgery, it is also known that a significant systemic inflammatory response is mounted in patients who undergo conventional CPB. This inflammatory response is a combined effect of 1) the placement of required tubes and lines for connection with the heart/lung machine, 2) hemodilution, and 3) hypothermia. In this study, we will measure levels of tissue inflammation through the use of specialized laboratory tests (C Reactive Protein, C5 complement activation and Interleukin 6), and we will correlate these inflammation levels to the three different cardiopulmonary bypass options. It is our hypothesis that MECC will provide the stable operating environment of conventional CPB and the patient benefits of less blood loss, decreased transfusion rate, and decreased inflammation levels seen in patients with OPCAB.

Statistical Analysis: Multivariable regression models will be used to investigate the association of the MECC pump, conventional CPB versus off-pump with the outcomes controlling for risk factors recognized by the STS associated with post-CABG adverse outcomes) and other clinical and non-clinical factors. The association of each outcome of interest with MECC versus conventional CPB and MECC versus off-pump will be estimated with 95% confidence intervals (CIs). With a cohort of 102 patients (34 in each of three study groups) we will have over 80% power to detect a 71% relative reduction (30% absolute difference) in transfusion rate among CABG patients using a MECC pump as compared to conventional pump patients assuming that 42% of patients undergoing CABG with conventional pump require a transfusion

ELIGIBILITY:
Inclusion Criteria:

-Males and females at least 18 years of age undergoing CABG surgery who are suitable candidates cardiopulmonary bypass.

Exclusion Criteria:

* Candidate requires emergency surgery.
* Previous cardiac surgery.
* Plans for concomitant cardiac valve surgery. (Note: concomitant vein isolation is permissible).
* Pregnant or intends to become pregnant during the study.
* Candidate is unable or unwilling to provide informed consent participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital facility
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To compare blood loss and PRBC transfusions for MECC, OPCAB, and conventional CPB in patients undergoing primary CABG surgery. | 12 months

SECONDARY OUTCOMES:
To assess survival and readmission rates 30 days post discharge. | 1 year
  Description: Through interview and medical record review subjects will be assessed 30 days post discharge for readmissions, adverse events and survival
To assess and compare levels of tissue inflammation using biomarkers. | 1 year
  Blood samples collected at five timepoints preop, intraop and postoperatively will be evaluated for C-Reactive Protein, C5 Complement Activation and IL-6 levels and compared among the 3 groups.
To assess and compare levels of tissue inflammation using genomic mapping. | 1 year
  Compare blood levels of inflammation by completeing genomic mapping using micrarray technology
To identify a definition of a genomic signature of inflammation that predicts best outcomes in using CECC, MECC, and off-pump for CABG surgery. | 1 year
To use results of the trial to develop a a future large scale trial. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, Principal Investigator — The Heart Hospital at Baylor Plano
Locations (1):
- The Heart Hospital at Baylor Plano, Plano, Texas, United States